CLINICAL TRIAL: NCT04951284
Title: A Study to Evaluate the Ability of Speech- and Language-based Digital Biomarkers to Detect and Characterise Prodromal and Preclinical Alzheimer's Disease in a Clinical Setting - AMYPRED-US FUTURE Extension Study.
Brief Title: Amyloid Prediction in Early Stage Alzheimer's Disease Through Speech Phenotyping - FUTURE Extension
Acronym: FUTURE-US
Status: Terminated | Type: Observational
Why Stopped: Study only continued to 2 year follow-up.
Sponsor: Novoic Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: NOV-0110-1
Record Dates: First submitted 2021-06-17; First posted 2021-07-06 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Alzheimer Disease; Preclinical Alzheimer's Disease; Prodromal Alzheimer's Disease; Alzheimer's Disease (Incl Subtypes); Mild Cognitive Impairment
Keywords: Alzheimer's disease; Preclinical Alzheimer's disease; Prodromal Alzheimer's disease; Mild Cognitive Impairment; Normal Cognition; Amyloid; Speech; Acoustic; Language; Linguistic; Machine Learning; Artificial Intelligence
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Speech; Language

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Arm 1: MCI amyloid positive: * Meet the National Institute of Aging - Alzheimer's Association (NIA-AA) core clinical criteria (2011) for MCI due to Alzheimer's
  * Positive amyloid PET or amyloid CSF status.
  * MMSE 23-30 (inclusive)
- Arm 2: MCI amyloid negative: * Non-AD Mild Cognitive Impairment (MCI)
  * Negative amyloid PET or amyloid CSF status.
  * MMSE 23-30 (inclusive)
- Arm 3: CN amyloid positive: * Absence of a diagnosis of cognitive disorder and/or subjectively reported cognitive decline
  * Positive amyloid PET or amyloid CSF status.
  * MMSE 26-30 (inclusive)
- Arm 4: CN amyloid negative: * Absence of a diagnosis of cognitive disorder and/or subjectively reported cognitive decline
  * Negative amyloid PET or amyloid CSF status.
  * MMSE 26-30 (inclusive)

SUMMARY:
The primary objective of the study is to evaluate whether a set of algorithms analysing acoustic and linguistic patterns of speech, can predict change in Preclinical Alzheimer's Clinical Composite with semantic processing (PACC5) between baseline and +12 month follow up across all four Arms, as measured by the coefficient of individual agreement (CIA) between the change in PACC5 and the corresponding regression model, trained on baseline speech data to predict it. Secondary objectives include (1) evaluating whether similar algorithms can predict change in PACC5 between baseline and +12 month follow up in the cognitively normal (CN) and MCI populations separately; (2) evaluating whether similar algorithms trained to regress against PACC5 scores at baseline, still regress significantly against PACC5 scores at +12 month follow-up, as measured by the coefficient of individual agreement (CIA) between the PACC5 composite at +12 months and the regression model, trained on baseline speech data to predict PACC5 scores at baseline; (3) evaluating whether similar algorithms can classify converters vs non-converters in the cognitively normal Arms (Arm 3 + 4), and fast vs slow decliners in the MCI Arms (Arm 1 + 2), as measured by the Area Under the Curve (AUC) of the receiver operating characteristic curve, sensitivity, specificity and Cohen's kappa of the corresponding binary classifiers. Secondary objectives include the objectives above, but using time points of +24 months and +36 months; and finally to evaluate whether the model performance for the objectives and outcomes above improved if the model has access to speech data at 1 week, 1 month, and 3 month timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are fully eligible for and have completed the AMYPRED-US (Amyloid Prediction in early stage Alzheimer's disease from acoustic and linguistic patterns of speech) study.

(See https://clinicaltrials.gov/ct2/show/NCT04928976)

- Subject consents to take part in FUTURE extension study.

Exclusion Criteria:

* Subject hasn't completed the full visit day in the AMYPRED-US study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be identified from participants of the AMYPRED-US study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
The agreement between the change in the PACC5 composite between baseline and +12 months and the corresponding regression model, trained on baseline speech data, predicting in all four Arms, as measured by the coefficient of individual agreement (CIA). | 12 months

SECONDARY OUTCOMES:
The agreement between the change in the PACC5 composite between baseline and +24 months and the corresponding regression model, trained on baseline speech data, predicting in all four Arms, as measured by the coefficient of individual agreement (CIA). | 24 months
The agreement between the change in the PACC5 composite between baseline and +36 months and the corresponding regression model, trained on baseline speech data, predicting in all four Arms, as measured by the coefficient of individual agreement (CIA). | 36 months
The agreement between the change in the PACC5 composite between baseline and +12 months and the corresponding regression model, trained on baseline speech data, to predict it in the CN Arms (Arms 3 and 4), as measured by the CIA. | 12 months
The agreement between the change in the PACC5 composite between baseline and +24 months and the corresponding regression model, trained on baseline speech data, to predict it in the CN Arms (Arms 3 and 4), as measured by the CIA. | 24 months
The agreement between the change in the PACC5 composite between baseline and +36 months and the corresponding regression model, trained on baseline speech data, predicting it in the MCI Arms (Arms 1 and 2), as measured by the CIA. | 36 months
The agreement between the PACC5 composite at +12 months and the corresponding regression model, trained on baseline speech data, predicting in all four Arms based on +12 month speech data, as measured by the coefficient of individual agreement (CIA). | 12 months
The agreement between the PACC5 composite at +24 months and the corresponding regression model, trained on baseline speech data, predicting in all four Arms based on +12 month speech data, as measured by the coefficient of individual agreement (CIA). | 24 months
The agreement between the PACC5 composite at +36 months and the corresponding regression model, trained on baseline speech data, predicting in all four Arms based on +12 month speech data, as measured by the coefficient of individual agreement (CIA). | 36 months
The agreement between the PACC5 composite and the corresponding regression model, trained on baseline speech data and +12 month speech data, as measured by the coefficient of individual agreement (CIA). | 12 months
The agreement between the PACC5 composite and the corresponding regression model, trained on baseline speech data and +24 month speech data, as measured by the coefficient of individual agreement (CIA). | 24 months
The agreement between the PACC5 composite and the corresponding regression model, trained on baseline speech data and +36 month speech data, as measured by the coefficient of individual agreement (CIA). | 36 months
The AUC of the binary classifier distinguishing between converters vs non-converters in the cognitively normal (CN) Arms (Arms 3 and 4); converters defined as having a CDR Global score of 0.5 or more at +12 months. | 12 months
The AUC of the binary classifier distinguishing between converters vs non-converters in the cognitively normal (CN) Arms (Arms 3 and 4); converters defined as having a CDR Global score of 0.5 or more at +24 months. | 24 months
The AUC of the binary classifier distinguishing between converters vs non-converters in the cognitively normal (CN) Arms (Arms 3 and 4); converters defined as having a CDR Global score of 0.5 or more at +36 months. | 36 months
The sensitivity of the binary classifier distinguishing between converters vs non-converters in the cognitively normal (CN) Arms (Arms 3 and 4); converters defined as having a CDR Global score of 0.5 or more at +12 months. | 12 months
The sensitivity of the binary classifier distinguishing between converters vs non-converters in the cognitively normal (CN) Arms (Arms 3 and 4); converters defined as having a CDR Global score of 0.5 or more at +24 months. | 24 months
The sensitivity of the binary classifier distinguishing between converters vs non-converters in the cognitively normal (CN) Arms (Arms 3 and 4); converters defined as having a CDR Global score of 0.5 or more at +36 months. | 36 months
The specificity of the binary classifier distinguishing between converters vs non-converters in the cognitively normal (CN) Arms (Arms 3 and 4); converters defined as having a CDR Global score of 0.5 or more at +12 months. | 12 months
The specificity of the binary classifier distinguishing between converters vs non-converters in the cognitively normal (CN) Arms (Arms 3 and 4); converters defined as having a CDR Global score of 0.5 or more at +24 months. | 24 months
The specificity of the binary classifier distinguishing between converters vs non-converters in the cognitively normal (CN) Arms (Arms 3 and 4); converters defined as having a CDR Global score of 0.5 or more at +36 months. | 36 months
The Cohen's kappa of the binary classifier distinguishing between converters vs non-converters in the cognitively normal (CN) Arms (Arms 3 and 4); converters defined as having a CDR Global score of 0.5 or more at +12 months. | 12 months
The Cohen's kappa of the binary classifier distinguishing between converters vs non-converters in the cognitively normal (CN) Arms (Arms 3 and 4); converters defined as having a CDR Global score of 0.5 or more at +24 months. | 24 months
The Cohen's kappa of the binary classifier distinguishing between converters vs non-converters in the cognitively normal (CN) Arms (Arms 3 and 4); converters defined as having a CDR Global score of 0.5 or more at +36 months. | 36 months
The AUC of the binary classifier distinguishing between fast decliners vs slow decliners in the MCI Arms (Arms 1 and 2) at +12 months. | 12 months
The AUC of the binary classifier distinguishing between fast decliners vs slow decliners in the MCI Arms (Arms 1 and 2) at +24 months. | 24 months
The AUC of the binary classifier distinguishing between fast decliners vs slow decliners in the MCI Arms (Arms 1 and 2) at +36 months. | 36 months
The sensitivity of the binary classifier distinguishing between fast decliners vs slow decliners in the MCI Arms (Arms 1 and 2) at +12 months. | 12 months
The sensitivity of the binary classifier distinguishing between fast decliners vs slow decliners in the MCI Arms (Arms 1 and 2) at +24 months. | 24 months
The sensitivity of the binary classifier distinguishing between fast decliners vs slow decliners in the MCI Arms (Arms 1 and 2) at +36 months. | 36 months
The specificity of the binary classifier distinguishing between fast decliners vs slow decliners in the MCI Arms (Arms 1 and 2) at +12 months. | 12 months
The specificity of the binary classifier distinguishing between fast decliners vs slow decliners in the MCI Arms (Arms 1 and 2) at +24 months. | 24 months
The specificity of the binary classifier distinguishing between fast decliners vs slow decliners in the MCI Arms (Arms 1 and 2) at +36 months. | 36 months
The Cohen's kappa of the binary classifier distinguishing between fast decliners vs slow decliners in the MCI Arms (Arms 1 and 2) at +12 months. | 12 months
The Cohen's kappa of the binary classifier distinguishing between fast decliners vs slow decliners in the MCI Arms (Arms 1 and 2) at +24 months. | 24 months
The Cohen's kappa of the binary classifier distinguishing between fast decliners vs slow decliners in the MCI Arms (Arms 1 and 2) at +36 months. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Emil Fristed, MSc, Principal Investigator — Novoic Ltd
Locations (1):
- Syrentis Clinical Research, Santa Ana, California, United States

IPD SHARING:
Plan to Share IPD: Undecided